CLINICAL TRIAL: NCT04559958
Title: Tongue Inspection and Diagnosis for Chronic Kidney Disease: Protocol for a Cross-sectional, Case-controlled Observational Study
Brief Title: Tongue Diagnosis in Chronic Kidney Disease
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CMPRG8H0691
Record Dates: First submitted 2020-09-14; First posted 2020-09-23 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2018-09

CONDITIONS: Chronic Kidney Diseases
Keywords: Chronic kidney diseases; Automatic tongue diagnosis system; Traditional Chinese medicine
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- non-dialysis CKD group: Participants with estimated glomerular ﬁltration rate (eGFR) <60 mL/min/1.73 m2 more than three months and without regular dialysis will be enrolled in non-dialysis CKD group.
  Interventions: Diagnostic Test: tongue image
- ESRD group: Participants with eGFR ≤15 mL/min/1.73 m2 and underwent regular dialysis will be recruited in ESRD group.
  Interventions: Diagnostic Test: tongue image
- control group: Participants with eGFR ≧60 mL/min/1.73 m2 and without evidence of kidney damage such as albuminuria or abnormal findings on renal imaging will be enrolled in control group.
  Interventions: Diagnostic Test: tongue image

INTERVENTIONS:
Diagnostic Test: tongue image — capture tongue images by Automatic Tongue Diagnosis System

SUMMARY:
The Automatic Tongue Diagnosis System (ATDS) was developed to capture tongue images and extract features reliably to assist the diagnosis of traditional chinese medicine (TCM) practitioners.This project will employ the ATDS verified to extract the tongue features of patients with chronic kidney disease. A TCM indices derived through the non-intrusive tongue diagnosis procedure can provide valuable information for clinical doctors to analyze the current status of a patient and dynamically schedule a treatment plan, facilitating early detection and diagnosis of chronic kidney disease.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is a global financial and medical burden, because its high morbidity and mortality. Tongue diagnosis is an important diagnostic tool in traditional Chinese medicine. However, tongue diagnosis often biased by subjective judgements and environmental factors. The automatic tongue diagnosis system can noninvasively capture tongue images, automatically correct any lighting and color deviation and analyze tongue manifestations.

This protocol is a cross-sectional, case-controlled observational study investigating the tongue features of non-dialysis CKD and end-stage renal disease patients by using the noninvasive ATDS. CKD patients who meets inclusion and exclusion criteria will be enrolled. Participants will be divided into 3 groups according to their renal function and accept dialysis or not, including a non-dialysis CKD group, end stage renal disease (ESRD) group and control group. Tongue images will be captured and 9 tongue features including tongue shape, tongue color, fur thickness, fur color, saliva, tongue fissure, ecchymosis, tooth mark, and red dots will be extracted and analyzed by ATDS.

This protocol aims to apply noninvasive ATDS to analyze tongue features of CKD patients.

ELIGIBILITY:
Inclusion Criteria:

The patients will be included if they meet the following criteria:

1. age over 20 years old
2. The person who volunteered to participate this research and signed the agreement of institutional review board.

Exclusion Criteria:

1. Pregnant women
2. Patients with acute infection
3. The person who has cancer with brain metastasis and present with cognitive dysfunction such as dementia or delirium
4. unable to protrude the tongue stably
5. Patients with risk of temporomandibular joint dislocation
6. Those who did not sign the agreement of institutional review board

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with chronic kidney diseases
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Tongue features | day 1
  diagnosed by the Automatic Tongue Diagnosis System (ATDS)

SECONDARY OUTCOMES:
serum blood urea nitrogen (BUN) | day 1
  renal function test
serum creatinine | day 1
  renal function test
eGFR | day 1
  eGFR is calculated by using the Modiﬁcation of Diet in Renal Disease Study equation
hemoglobin | day 1
  evaluate anemia

CONTACTS AND LOCATIONS:
Overall Officials: yu-chiang hung, Ph.D., Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tsai MH, Hsu CY, Lin MY, Yen MF, Chen HH, Chiu YH, Hwang SJ. Incidence, Prevalence, and Duration of Chronic Kidney Disease in Taiwan: Results from a Community-Based Screening Program of 106,094 Individuals. Nephron. 2018;140(3):175-184. doi: 10.1159/000491708. Epub 2018 Aug 23. PMID 30138926
- [Result] Hsu PC, Wu HK, Huang YC, Chang HH, Lee TC, Chen YP, Chiang JY, Lo LC. The tongue features associated with type 2 diabetes mellitus. Medicine (Baltimore). 2019 May;98(19):e15567. doi: 10.1097/MD.0000000000015567. PMID 31083226
- [Result] Lee TC, Lo LC, Wu FC. Traditional Chinese Medicine for Metabolic Syndrome via TCM Pattern Differentiation: Tongue Diagnosis for Predictor. Evid Based Complement Alternat Med. 2016;2016:1971295. doi: 10.1155/2016/1971295. Epub 2016 May 25. PMID 27313640
- [Result] Lo LC, Cheng TL, Chen YJ, Natsagdorj S, Chiang JY. TCM tongue diagnosis index of early-stage breast cancer. Complement Ther Med. 2015 Oct;23(5):705-13. doi: 10.1016/j.ctim.2015.07.001. Epub 2015 Jul 10. PMID 26365451
- [Result] Kim J, Han G, Ko SJ, Nam DH, Park JW, Ryu B, Kim J. Tongue diagnosis system for quantitative assessment of tongue coating in patients with functional dyspepsia: a clinical trial. J Ethnopharmacol. 2014 Aug 8;155(1):709-13. doi: 10.1016/j.jep.2014.06.010. Epub 2014 Jun 13. PMID 24933221
- [Result] Levin A, Stevens PE. Summary of KDIGO 2012 CKD Guideline: behind the scenes, need for guidance, and a framework for moving forward. Kidney Int. 2014 Jan;85(1):49-61. doi: 10.1038/ki.2013.444. Epub 2013 Nov 27. PMID 24284513
- [Result] Levey AS, Bosch JP, Lewis JB, Greene T, Rogers N, Roth D. A more accurate method to estimate glomerular filtration rate from serum creatinine: a new prediction equation. Modification of Diet in Renal Disease Study Group. Ann Intern Med. 1999 Mar 16;130(6):461-70. doi: 10.7326/0003-4819-130-6-199903160-00002. PMID 10075613
- [Result] Drawz P, Rahman M. Chronic kidney disease. Ann Intern Med. 2015 Jun 2;162(11):ITC1-16. doi: 10.7326/AITC201506020. PMID 26030647
- [Result] Meyer TW, Hostetter TH. Uremia. N Engl J Med. 2007 Sep 27;357(13):1316-25. doi: 10.1056/NEJMra071313. No abstract available. PMID 17898101
- [Result] Almeras C, Argiles A. The general picture of uremia. Semin Dial. 2009 Jul-Aug;22(4):329-33. doi: 10.1111/j.1525-139X.2009.00575.x. PMID 19708976
- [Result] Zhong Y, Deng Y, Chen Y, Chuang PY, Cijiang He J. Therapeutic use of traditional Chinese herbal medications for chronic kidney diseases. Kidney Int. 2013 Dec;84(6):1108-18. doi: 10.1038/ki.2013.276. Epub 2013 Jul 17. PMID 23868014
- [Result] Zhong Y, Menon MC, Deng Y, Chen Y, He JC. Recent Advances in Traditional Chinese Medicine for Kidney Disease. Am J Kidney Dis. 2015 Sep;66(3):513-22. doi: 10.1053/j.ajkd.2015.04.013. Epub 2015 May 23. PMID 26015275
- [Result] Xiong W, He FF, You RY, Xiong J, Wang YM, Zhang C, Meng XF, Su H. Acupuncture Application in Chronic Kidney Disease and its Potential Mechanisms. Am J Chin Med. 2018;46(6):1169-1185. doi: 10.1142/S0192415X18500611. PMID 30286626
- [Result] Tania MH, Lwin K, Hossain MA. Advances in automated tongue diagnosis techniques. Integr Med Res. 2019 Mar;8(1):42-56. doi: 10.1016/j.imr.2018.03.001. Epub 2018 Mar 8. PMID 30949431
- [Result] Liu Q, Yue XQ, Ling CQ. [Researches into the modernization of tongue diagnosis: in retrospect and prospect]. Zhong Xi Yi Jie He Xue Bao. 2003 May;1(1):66-70. doi: 10.3736/jcim20030128. Chinese. PMID 15339625
- [Result] Anastasi JK, Currie LM, Kim GH. Understanding diagnostic reasoning in TCM practice: tongue diagnosis. Altern Ther Health Med. 2009 May-Jun;15(3):18-28. PMID 19472861
- [Result] Jung CJ, Jeon YJ, Kim JY, Kim KH. Review on the current trends in tongue diagnosis systems. Integr Med Res. 2012 Dec;1(1):13-20. doi: 10.1016/j.imr.2012.09.001. Epub 2012 Oct 5. PMID 28664042
- [Result] Chiu CC. A novel approach based on computerized image analysis for traditional Chinese medical diagnosis of the tongue. Comput Methods Programs Biomed. 2000 Feb;61(2):77-89. doi: 10.1016/s0169-2607(99)00031-0. PMID 10661393